CLINICAL TRIAL: NCT06980025
Title: A Dose Escalation Study of Low Dose Aspirin for the Prevention of Recurrent Preterm Birth
Brief Title: Aspirin Dose Escalation for the Prevention of Recurrent Preterm Delivery Trial
Acronym: ADEPT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Columbia University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD1036801-ADEPT; U01HD109332 (NIH); U24HD036801 (NIH)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Preterm Delivery; Obstetrical Complications
Keywords: Preterm Delivery; Stillbirth; Maternal Morbidity; Neonatal Morbidity; Prevention
MeSH Terms: conditions — Premature Birth; Stillbirth | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized between 10 weeks, 0 days gestation and 15 weeks, 6 days gestation to either aspirin 162 mg or aspirin 81 mg daily and continue the study intervention through 36 weeks, 6 days gestation. Randomization will be stratified by clinical site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study intervention is packaged and shipped from the central distribution center to the clinical sites. Participants, clinical staff, and clinical site investigators and research staff are masked to the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 162mg Aspirin Daily (Experimental): One 81mg capsule of aspirin daily through 36 weeks 6 days gestation.
  Interventions: Drug: 162mg Aspirin
- 81mg Aspirin Daily (Experimental): Two 81mg capsules of aspirin daily through 36 weeks 6 days gestation.
  Interventions: Drug: 81mg Aspirin

INTERVENTIONS:
Drug: 162mg Aspirin — Two 81mg aspirin tablets in an over-encapsulated capsule filled with microcrystalline cellulose.
  Study intervention will be packaged into bottles (35 capsules per bottle).
  Arms: 162mg Aspirin Daily
Drug: 81mg Aspirin — One 81mg aspirin tablet in an over-encapsulated capsule filled with microcrystalline cellulose.
  Study intervention will be packaged into bottles (35 capsules per bottle).
  Arms: 81mg Aspirin Daily

SUMMARY:
This is a phase-III multi-center double-blind randomized clinical trial of 1,800 individuals with a history of prior preterm birth at less than 35 weeks gestation who are randomized to either 162 mg aspirin or 81 mg aspirin daily. The study drug will be initiated between 10 and 15 weeks gestation and continued through 36 weeks, 6 days gestation. The primary endpoint is recurrent preterm delivery or fetal death prior to 35 weeks, 0 days gestation.

DETAILED DESCRIPTION:
This is a phase-III multi-center double-blind randomized clinical trial of 1,800 individuals with a history of prior preterm birth at less than 35 weeks gestation who are randomized to either 162 mg aspirin or 81 mg aspirin daily.

The primary objective is to assess the efficacy of daily 162 mg of aspirin compared to 81 mg aspirin in reducing recurrent preterm delivery or fetal death before 35 weeks, 0 days gestation in individuals with a proximal birth between 20 weeks, 0 days and 34 weeks, 6 days gestation with spontaneous preterm delivery (sPTB), ischemic placental disease (IPD), or stillbirth. Ischemic placental disease includes small for gestational age, preeclampsia, or placental abruption.

The secondary objective is to assess the efficacy of daily 162 mg of aspirin compared to 81 mg aspirin in reducing ischemic placental disease in individuals with a proximal birth between 20 weeks, 0 days and 34 weeks, 6 days gestation with sPTB, IPD, or stillbirth.

Tertiary /Exploratory objectives are 1) to assess the efficacy of daily 162 mg of aspirin compared to 81 mg aspirin in reducing adverse maternal and neonatal outcomes, and 2) to assess maternal and neonatal safety in individuals with a proximal birth between 20 weeks, 0 days and 34 weeks, 6 days gestation with sPTB, IPD, or stillbirth.

Individuals will be randomized between 10 and 15 weeks gestation to either 162mg or 81mg of aspirin daily and continue the study intervention through 36 weeks, 6 days gestation. Participants will have monthly virtual or in-person visits through 37 weeks gestation to assess study intervention compliance, side effects, medication use, and unscheduled hospitalization. Maternal blood will be collected in a subset of the population. Research staff will abstract maternal and neonatal outcomes following delivery and discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* 14 years or older
* Singleton gestation. Twin gestation reduced to a singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 13 weeks 6 days project gestational age. Higher-order multifetal gestations reduced to singletons are not eligible.
* Gestational age at randomization between 10 weeks 0 days and 15 weeks 6 days based on clinical information and evaluation of the earliest ultrasound.
* Prior preterm birth between 20 weeks 0 days and 34 weeks 6 days with one of the following in the proximal birth reaching 20 weeks or greater:

  * Spontaneous preterm birth is defined as spontaneous preterm labor or premature rupture of membranes
  * Ischemic placental disease is defined as preeclampsia, small for gestational age, fetal growth restriction, or placental abruption, as defined clinically.
  * Stillbirth excluding those with known genetic disorders or major congenital anomalies.

Exclusion Criteria:

* Known allergy or hypersensitivity to aspirin or any medical condition where aspirin is contraindicated (e.g., history of peptic ulcer disease, nasal polyps, NSAID-induced asthma, history of gastrointestinal bleeding, known G6PD deficiency, severe hepatic dysfunction, bleeding disorders, and consumption of 3 or more alcoholic drinks per day)
* Taking other anticoagulants such as Heparin or Low-Molecular weight Heparin
* Thrombocytopenia defined as a platelet count defined as a platelet count <100,000 microliters
* Gastric bypass surgery, regardless of type
* Aspirin use >81 mg daily during the current pregnancy who are not willing or able to go through a 2-week washout before randomization.
* Known major Mullerian anomaly of the uterus (specifically bicornuate, unicornuate, or uterine septum not resected) due to increased risk of preterm delivery.
* Known fetal genetic disease or major malformations
* Fetal demise or planned termination of pregnancy. Selective reduction by 13 weeks 6 days gestation, from twins to singleton, is not an exclusion.
* Any fetal/maternal condition requiring invasive in-utero assessment or treatment, for example, significant red cell antigen sensitization or neonatal alloimmune thrombocytopenia.
* Patients with any of the following medical conditions because of increased risk for adverse pregnancy outcome or indicated preterm birth:

  * Treated hypertension requiring more than one agent
  * Chronic renal disease with baseline serum creatinine ≥1.5 mg/dL
  * Conditions treated with chronic oral glucocorticoid therapy (e.g., systemic lupus erythematosus)
  * Uncontrolled hyper- and hypothyroid disease
  * New York Heart Association (NYHA) stage II or greater cardiac disease
* Planned indicated delivery prior to 37 weeks.
* Participation in another interventional study that influences the primary outcome in this study (gestational age at delivery).
* Participation in this trial in a previous pregnancy.
* Delivery planned at a non-participating site

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrent preterm delivery or fetal death prior to 35 weeks 0 days gestation | Between randomization and 35 weeks, 0 days gestation (a period of up to 25 weeks)
  Number and rate of participants who experience a recurrent preterm delivery or fetal death before 35 weeks, 0 days gestation.

SECONDARY OUTCOMES:
Rate of ischemic placental disease | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants who experience ischemic placental disease (preeclampsia, small for gestational age <10th percentile, or placental abruption). Small for gestational age is defined by "A 2017 US reference for singleton birth weight percentiles using obstetric estimates of gestation" by Aris et. al (2019).

OTHER OUTCOMES:
Rate of recurrent preterm delivery or fetal death at <28 weeks | Between randomization and delivery (a period of up to 18 weeks)
  Number and rate of participants who experience a recurrent preterm delivery or fetal death at less than 28 weeks
Rate of recurrent preterm delivery or fetal death at <37 weeks | Between randomization and delivery (a period of up to 27 weeks)
  Number and rate of participants who experience a recurrent preterm delivery or fetal death at less than 37 weeks
Rate of ischemic placental disease with delivery prior to 28 weeks | Between randomization and delivery (a period of up to 18 weeks)
  Number and rate of participants who experience ischemic placental disease (preeclampsia, fetal growth restriction, or placental abruption) with delivery before 28 weeks gestation
Rate of ischemic placental disease with delivery prior to 35 weeks | Between randomization and delivery (a period of up to 25 weeks)
  Number and rate of participants who experience ischemic placental disease (preeclampsia, fetal growth restriction, or placental abruption) with delivery before 35 weeks gestation
Rate of Ischemic Placental Disease with Delivery Prior to 37 weeks | Between randomization and delivery (a period of up to 27 weeks)
  Number of participants who experience ischemic placental disease (preeclampsia, fetal growth restriction, or placental abruption) with delivery before 37 weeks gestation
Rate of preeclampsia | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants who experience preeclampsia
Rate of preeclampsia with severe features | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants who experience preeclampsia with severe features including HELLP syndrome and eclampsia
Rate of placental abruption | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants who experience placental abruption as defined clinically (not pathologically determined)
Number of emergency room visits or hospitalizations | Between randomization and delivery (a period of up to 32 weeks)
  Mean or median number of non-scheduled emergency room visits or hospitalizations
Number of days between randomization and delivery or fetal death | Between randomization and delivery (a period of up to 32 weeks)
  Mean or median number of days between randomization and delivery or fetal death
Rate of stillbirth | Between 20 weeks gestation and delivery (a period of up to 22 weeks)
  Number and rate of stillbirths defined as fetal deaths occurring on or after 20 weeks, 0 days gestation
Rate of small for gestational age at less than 5th percentile | At delivery
  Number and rate of neonates determined to be small for gestational age at less than the 5th percentile. Small for gestational age is defined by "A 2017 US reference for singleton birth weight percentiles using obstetric estimates of gestation" by Aris et. al (2019).
Rate of small for gestational age at less than 10th Percentile | At delivery
  Number of neonates determined to be small for gestational age at less than the 10th percentile. Small for gestational age is defined by "A 2017 US reference for singleton birth weight percentiles using obstetric estimates of gestation" by Aris et. al (2019).
Rate of neonatal death | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonatal deaths
Rate of neonatal intensive care unit (NICU) admission | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates admitted to the neonatal intensive care unit (NICU)
Neonatal Length of Hospital Stay | Between delivery and hospital discharge (a period of up to 120 days)
  Mean or median number of days neonates stayed hospitalized
Rate of neonatal ventilator or continuous positive airway pressure (CPAP use | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates who needed ventilator or continuous positive airway pressure (CPAP) use
Rate of neonatal oxygen use | Between delivery and 72 hours post birth
  Number and rate of neonates who used oxygen for at least 4 continuous hours in the first 72 hours from birth
Rate of neonatal seizure | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates who experienced seizures requiring treatment
Rate of neonatal hyperbilirubinemia | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates who experienced hyperbilirubinemia requiring treatment
Rate of neonatal infectious morbidity | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates who experienced neonatal infectious morbidity defined as any one of the following: suspected sepsis, early onset sepsis, late onset sepsis, or pneumonia
Rate of perinatal composite outcome | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates with the perinatal composite outcome defined as any of the following:
  * Fetal or neonatal death
  * Bronchopulmonary dysplasia (BPD) grade 3 or higher
  * Intraventricular hemorrhage (IVH) grades 3 or 4
  * Necrotizing enterocolitis (NEC) proven - Bell Stage 2A or greater
  * Periventricular leukomalacia (PVL)
  * Retinopathy of prematurity (ROP) stage III-V
  * Proven sepsis (early or late)
Rate of minor bleeding | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants who reported minor bleeding defined as any of the following: vaginal spotting, gum, or nasal bleeding not requiring surgical coagulation/ packing.
Rate of thrombocytopenia | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants with thrombocytopenia defined as a platelet count < 100k
Rate of aspirin allergy | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants that report an allergic reaction to aspirin
Rate of gastric ulcer disease | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants that report active gastric ulcer disease that is not responsive to common therapies
Rate of persistent epistaxis | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants that report persistent epistaxis (nosebleeds) defined as prolonged nosebleeds that last for more than 15 minutes or occur more than once a week, or require medical intervention.
Rate of clinically meaningful bleeding | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants that report clinically meaningful bleeding defined as any of the following: abruption, hemoptysis (coughing up blood or bloody mucus), nasal bleeding requiring coagulation or packing
Estimated blood loss | Delivery
  Mean or median estimated blood loss during delivery
Rate of estimated blood loss greater than 1000ml | Delivery
  Number and rate of participants that have an estimated blood loss during delivery greater than 1000ml
Rate of transfusion of packed red blood cells | Between delivery admission and hospital discharge (a period of up to 120 days)
  Number and rate of participants that have a transfusion of packed red blood cells
Rate of cesarean hysterectomy | Delivery
  Number and rate of participants who had a cesarean hysterectomy
Rate of intensive care unit (ICU) admission | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants admitted to the intensive care unit (ICU)
Rate of intracranial hemorrhage | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants who experienced an intracranial hemorrhage
Rate of congenital malformation | Between randomization and hospital discharge (a period of up to 49 weeks)
  Number and rate of congenital malformation and premature narrowing or closure of the ductus arteriosus
Rate of oligohydramnios | Between randomization and delivery (a period of up to 32 weeks)
  Number and rate of participants with clinically-defined oligohydramnios
Rate of neonatal primary pulmonary hypertension | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates with primary pulmonary hypertension
Rate of neonatal intracranial hemorrhage | Between delivery and hospital discharge (a period of up to 120 days)
  Number and rate of neonates with perinatal intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Clifton, PhD, Principal Investigator — The George Washington University Biostatistics Center; Matthew K Hoffman, MD, MPH, Principal Investigator — ChristianaCare Center for Women & Children's Health Research; Uma M Reddy, MD, MPH, Principal Investigator — Columbia University; Cande Ananth, PhD, MPH, Principal Investigator — Robert Wood Johnson Medical School - Rutgers Health
Locations (14):
- United States (14):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Regents of the University of California San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via NICHD DASH in accordance with NIH policy.
Supporting Information: Study Protocol, ICF